CLINICAL TRIAL: NCT00994448
Title: Pilot Trial of Bupropion Versus Placebo for Methamphetamine Abuse in Adolescents
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); Behavioral Health Services, Inc. (Industry)
Responsible Party: Principal Investigator, Keith Heinzerling, Assistant Clinical Professor, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1R21DA026513 (NIH)
Record Dates: First submitted 2009-10-13; First posted 2009-10-14 (Estimated); Results first posted 2013-04-04 (Estimated); Last update posted 2013-04-04 (Estimated); Status verified 2013-02

CONDITIONS: Adolescent Methamphetamine Abuse
Keywords: Adolescents; Methamphetamine abuse; Bupropion; Addiction; Pharmacotherapy; Cognitive Behavioral Therapy; Contingency Management; Teens
MeSH Terms: conditions — Behavior, Addictive

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bupropion (Experimental)
  Interventions: Drug: Bupropion SR 150mg tabs
- Placebo (sugar pill) (Placebo Comparator)
  Interventions: Drug: Placebo tablets

INTERVENTIONS:
Drug: Bupropion SR 150mg tabs — Bupropion SR 150mg tabs (Zyban) twice daily
  Arms: Bupropion
Drug: Placebo tablets — One placebo tablet twice daily
  Arms: Placebo (sugar pill)

SUMMARY:
Dr Keith Heinzerling, who is a doctor at UCLA, is doing a research study with Behavioral Health Services in the Lincoln Heights neighborhood of Los Angeles to find out if a medication called bupropion can help adolescents (age 14-21) reduce or stop using methamphetamine. Bupropion is a drug that is already on the market, which means it has been approved by the FDA, but it has not been approved to treat methamphetamine abuse. What the study is trying to find out is if bupropion helps people to stop using methamphetamine. The study lasts up to 14 weeks and involves visits to the BHS clinic in Lincoln Heights twice a week. The first two weeks involve completion of questionnaires and assessments, including a physical exam, a blood test, EKG (a test that checks for problems with the electrical activity of a person's heart), and a psychological interview, to see if you are eligible for the study. If you are eligible, then you will be assigned by chance to take either the bupropion pills or placebo pills, which are pills that look the same, but contain no medication. This type of study is called a "double blind study" because neither you nor any of the study staff will know which medication you are taking. During the 8 weeks of taking the pills, you'll visit the clinic to complete additional questionnaires and assessments, to provide urine samples for testing for methamphetamine, and for once a week drug abuse counseling. At the end of your treatment, you'll have another physical exam including blood tests and the same test on your heart and then we'll ask you to come to the clinic once a week for four weeks for follow-up assessments. You'll be compensated for time spent doing research activities and for returning empty medication packages. The total compensation possible is $332 in gift cards for places such as Target, iTunes, groceries, and gas.

Your participation in the study is voluntary and deciding not to participate or deciding to stop participating at any time during the study is okay.

ELIGIBILITY:
Inclusion Criteria:

1. age 14 years to 21 years of age, inclusive;
2. meet DSM-IV criteria for methamphetamine abuse or dependence as determined by the K-SADS-PL;
3. seeking treatment for MA problems;
4. report MA use on 18 or fewer of the past 30 days at baseline;
5. willing and able to comply with study procedures;
6. willing and able to provide informed assent (for youth <18 yr) or consent (for youth ≥18 yr) and parents willing to provide informed consent (for youth <18) to participate in the project; and
7. able to complete study assessments in English due to the lack of some measures in Spanish;
8. if female, not pregnant or lactating and willing to use an acceptable method of barrier birth control (e.g. condoms) during the trial.

Exclusion Criteria:

1. have a medical condition that, in the study physician's judgment, may interfere with safe study participation (e.g., active TB, unstable cardiac, renal, or liver disease, unstable diabetes);
2. have a current neurological disorder (e.g., organic brain disease, dementia) or major psychiatric disorder not due to substance abuse (e.g., schizophrenia, bipolar disorder) as assessed by the K-SADS-PL other than attention deficit-hyperactivity disorder (see below) or a medical history which would make study agent compliance difficult or which would compromise informed consent, or history of suicide attempts in the past year and/or current serious suicidal intention or plan as assessed by the K-SADS-PL;
3. currently taking bupropion for depression, smoking cessation or OCD within 30 days of baseline;
4. taking any prescription medication for ADHD;
5. currently on prescription medication that is contraindicated for use with bupropion;
6. have current dependence on cocaine, opiates, alcohol, or benzodiazepines as defined by DSM-IV-TR;
7. have a self-reported history of a seizure disorder or serious closed head injury;
8. have a medical condition (such as serious head injury) that is associated with increased risk of seizures or on a medication that lowers the seizure threshold;
9. have a current or past history of anorexia or bulimia;
10. body weight less than 50kgs;
11. have current hypertension uncontrolled by medication;
12. have a history of sensitivity to bupropion; and
13. any other circumstances that, in the opinion of the investigators, would compromise participant safety.

Ages: 14 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 19 (Actual)
Dates: Start 2009-10; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Keith Heinzerling, MD, MPH, Principal Investigator — UCLA Department of Family Medicine
Locations (1):
- Behavioral Health Services- Lincoln Heights Family Recovery Center, Los Angeles, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: substance abuse clinic, community outreach
Pre-assignment Details: Reasons for not being randomized were: withdrew voluntarily (4), failed to complete assessments (2), psychiatric disorder (2), weight < 50 kg (2), alcohol dependent (1), and incarcerated (1).
Groups:
- Bupropion: Bupropion SR 150 mg twice a day
- Placebo (Sugar Pill): Matching placebo tablets twice a day
Period: Overall Study
Arm/Group | Bupropion | Placebo (Sugar Pill)
Started | 12 | 7
Completed | 4 | 5
Not Completed | 8 | 2
Not completed — Adverse Event | 1 | 0
Not completed — Lost to Follow-up | 5 | 1
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bupropion | Placebo (Sugar Pill) | Total
Number analyzed (Participants) | 12 | 7 | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 7 | 4 | 11
  Between 18 and 65 years | 5 | 3 | 8
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 17.5 (1.6) | 17.7 (1.1) | 17.5 (1.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 3 | 10
  Male | 5 | 4 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 6 | 17
  Not Hispanic or Latino | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 0 | 0 | 0
  White | 12 | 6 | 18
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 12 | 7 | 19

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of Retaining Adolescents in Trial
Description: the mean retention for participants is used to assess feasibility of retaining adolescents in the trial (completion = 56 days or 8 weeks)
Time Frame: 8 weeks
Population: mean days retained in treatment for each grou[p
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Bupropion | Placebo (Sugar Pill)
Number analyzed (Participants) | 12 | 7
days | 33.3 (21.2) | 49.3 (9.8)
Statistical Analysis 1: Comparison: Bupropion vs Placebo (Sugar Pill); t test for mean of days retained in the bupropion versus placebo groups; Test type: Superiority or Other; p = 0.08, t-test, 2 sided; Mean Difference (Net) = 16.3, 95% CI 2-sided [1.8 to 34.3], Standard Error of Mean 8.6

ADVERSE EVENTS:
Arm/Group | Bupropion | Placebo (Sugar Pill)
Serious Adverse Events (participants affected / at risk) | 1/12 | 0/7
Other Adverse Events (participants affected / at risk) | 9/12 | 4/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bupropion (N=12) | Placebo (Sugar Pill) (N=7)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bupropion (N=12) | Placebo (Sugar Pill) (N=7)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Flu symptoms (Infections and infestations) | 2 (2) | 0 (0)
Upper Respiratory Infection (Infections and infestations) | 1 (1) | 1 (1)
Blurry Vision (Eye disorders) | 0 (0) | 1 (1)
Cold Sore (Infections and infestations) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Meth cravings (Psychiatric disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upset Stomach (Gastrointestinal disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Study was not powered or designed to determine if bupropion is more effective than placebo for treating methamphetamine dependence. Only for pilot testing procedures for a clinical trial in methamphetamine abusing adolescents.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No